CLINICAL TRIAL: NCT04649515
Title: Phase 3 Multi-Site, Randomised, Placebo Controlled, Double Blind, Single Dose Study of TY027 for Early Treatment of COVID-19
Brief Title: Efficacy and Safety of TY027, a Treatment for COVID-19, in Humans
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Low recruitment rate
Sponsor: Tychan Pte Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCT-301
Record Dates: First submitted 2020-11-26; First posted 2020-12-02 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Coronavirus Disease-2019 (COVID-19)
Keywords: Coronavirus Disease-2019; COVID-19; SARS-CoV-2; Monoclonal Antibody; Infectious diseases; Phase 3 study; Singapore
MeSH Terms: conditions — COVID-19; Communicable Diseases | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: Participants are assigned to either treatment or placebo
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TY027 1,500 mg (Experimental): 1,500 mg of TY027 will be administered via IV infusion over a period of 30 minutes.
  Interventions: Biological: TY027
- TY027 2,000 mg (Experimental): 2,000 mg of TY027 will be administered via IV infusion over a period of 30 minutes.
  Interventions: Biological: TY027
- Placebo (Placebo Comparator): Placebo will be administered via IV infusion over a period of 30 minutes.
  Interventions: Other: 0.9% saline

INTERVENTIONS:
Biological: TY027 — TY027 Injection, (100 mg/5 mL/Vial), SARS-CoV-2 Monoclonal Antibody (mAb) - 1,500 mg of TY027
  Arms: TY027 1,500 mg
Biological: TY027 — TY027 Injection, (100 mg/5 mL/Vial), SARS-CoV-2 Monoclonal Antibody (mAb) - 2,000 mg of TY027
  Arms: TY027 2,000 mg
Other: 0.9% saline — Placebo
  Arms: Placebo

SUMMARY:
The emergence & rapid spread of the coronavirus disease 2019 (COVID-19) since December 2019 across 188 countries globally has become a major public health crisis. COVID-19 was declared a pandemic by the World Health Organisation on 11 March 2020. To date, tens of millions of cases have been reported and over 3% of these cases have died. COVID-19 is an acute respiratory disease caused by the novel SARS-CoV-2 virus from the Betacoronavirus genus, just like SARS-CoV and MERS-CoV. SARS-CoV-2 is primarily transmitted person-to-person through respiratory droplets/close contact. Fomite transmission has also been shown as a transmission route. Common respiratory symptoms such as fever, sore throat, cough & shortness of breath, may appear 2 - 14 days after exposure. About 20% of infected cases progress to severe disease resulting in an estimated 2 - 5% mortality rate. With the unrelenting increase in cases being reported worldwide, there is thus an urgent need for therapeutics to be developed to treat disease & reduce further transmission in order to disrupt the ongoing pandemic.

To date, there are no specific proven antiviral treatment to prevent disease progression from mild to severe respiratory dysfunction among COVID-19 patients. Supportive care is recommended for symptom relief & for severe cases. Numerous vaccine candidates against SARS-CoV-2 are under development. Tychan's TY027, a fully engineered human IgG, is one of the first few biologics in the world, specifically targeting SARS-CoV-2, to enter human clinical trials. Preliminary data from our phase 1 healthy volunteer trial (SCT-001; ClinicalTrials.gov Identifier NCT04429529) reveals that TY027 is safe & well-tolerated up to 20 mg/kg tested. A total of 10 adverse events (AEs) were observed, all were of mild in intensity with none resulting in subject withdrawal from the study. There were no serious adverse events & no clinically relevant trends in mean clinical laboratory, physical examinations, vital signs or ECG results were observed. Pharmacokinetic profile of subjects across dose cohorts 1 - 4, up to Day 14, were comparable to those typical of human IgG1 antibody with serum concentrations declining in a biphasic manner. Exposure of TY027, based on Cmax, increased in a linear & generally dose proportional manner. It is anticipated that TY027, when administered to acutely infected COVID-19 patients, could reduce disease severity. It may potentially also be used as a prophylaxis against COVID-19 amongst high risk contacts.

DETAILED DESCRIPTION:
This is a Phase 3 Multi-Site, Randomised, Placebo Controlled, Double Blind, Single Dose Study of TY027 for Early Treatment of COVID-19.

Efficacy and safety of single dose IV infusion of TY027 in COVID-19 patients will be assessed.

A total of 1,305 COVID-19 patients will be enrolled. The first 15 patients will be randomised 1:1:1 to receive either (i) a single fixed dose of 1,500 mg TY027, (ii) a single fixed dose of 2,000 mg TY027 or (iii) Placebo (N = 5 per group) for initial safety assessment. This safety assessment will comprise the safety review of clinical signs, adverse events (AEs) and laboratory test results up to Day 3 post-dose.

Subsequent patients will be randomised 1:1 to receive either a single fixed dose of 2,000 mg TY027 (2,000 mg TY027 group) or Placebo (Placebo group) (N = 645 per group).

All patients will be inpatient for up to 7 days post-dosing and followed up on Days 14 and 28.

If a patient becomes clinically well enough for discharge before Day 7, at the discretion of attending physician, collection of subsequent events/parameters such as abbreviated physical examinations, vital signs, clinical laboratory assessments, pharmacodynamic assessment, biomarker assessment, disseminated intravascular coagulation assessment scheduled after discharge will no longer be feasbile. Conversely, if a patient was to be hospitalised beyond 7 days for medically indicated reasons, daily monitoring and medical assessment will continue, with any additional ad hoc sampling to be recorded as unscheduled visit(s).

Remote monitoring through a telephone or video call will be performed on days post-discharge as per originally scheduled in schedule of events, as well as on Day 14 while patients are serving their quarantine order or has been discharged home.

All discharged patients are to contact the Principal Investigator or the study team as soon as possible should they experience a worsening of their condition, or if they are admitted to hospital for COVID-19-related symptoms, before their Day 28 visit.

Final safety and efficacy analysis of all patients will be assessed at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic and RT-PCR confirmed COVID-19 within 6 days from symptom onset.
2. Has any one of the following factors associated with disease progression:

   1. Elevated lactate dehydrogenase (LDH)
   2. Elevated C reactive protein (CRP)
   3. Lymphocyte count below normal limit
   4. Age 40 and above
   5. History of well-controlled diabetes, hypertension, chronic obstructive lung disease or ischemic heart diseases
   6. Stable chronic renal disease
   7. History of asthma
3. Disease outcome score of 6, 7 or 8 based on the COVID Scale
4. Willing to comply with the requirements of the study protocol and attend scheduled study visits
5. Can give written informed consent approved by the Ethical Review Board governing the site

Exclusion Criteria:

1. Aged below 21 years old
2. Female who is pregnant or breast-feeding
3. With the following conditions, but not limited to:

   1. Known or suspected congenital or acquired immunodeficiency; or receipt of immunomodulation therapy such as anti-cancer chemotherapy or radiation therapy; or long-term systemic corticosteroid therapy defined as prednisone or equivalent for more than 2 consecutive weeks within the past 3 months
   2. Child-Pugh Class C chronic liver disease
   3. Renal insufficiency with an estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73m2 calculated by the CKD-EPI formula
   4. Suspected or confirmed active bacterial, fungal or mycobacterial infection
4. History of any allergic reaction to monoclonal antibodies
5. Currently enrolled in another COVID-19 investigational drug study
6. Previously enrolled in a COVID-19 investigational vaccine study
7. Any medical condition, which in the opinion of the Investigator, will compromise the safety of the patient

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-12-04 (Actual); Primary Completion 2022-03-04 (Actual); Study Completion 2022-03-04 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of a single dose intravenous (IV) infusion of TY027 in reducing disease progression, defined as progression to score 4 and below on COVID scale | Within the first 14 days
  Proportion of COVID-19 patients with disease progression, defined as progression to score 4 and below on the COVID Scale, within the first 14 days after a single dose IV infusion of TY027 as compared to placebo

SECONDARY OUTCOMES:
Rate of AEs (grade 3 and above) and SAEs in COVID-19 patients | 28 days
  Rate of AEs (grade 3 and above) and SAEs in COVID-19 patients after a single dose IV infusion of TY027 as compared to placebo
All cause mortality rate | 28 days
  All cause mortality rate by Day 28 in COVID-19 patients who receive a single dose IV infusion of TY027 as compared to placebo
Proportion of subjects in categories 4, 3, 2 and 1 of the COVID scale | Up to Day 28
  Proportion of subjects in categories 4, 3, 2 and 1 of the COVID scale at Day 7, Day 14 and Day 28
Number of days COVID-19 patients require supplemental oxygen, high flow oxygen, non-invasive and invasive mechanical ventilation (if applicable) | 28 days
  Number of days COVID-19 patients require supplemental oxygen, high flow oxygen, non-invasive and invasive mechanical ventilation (if applicable) after a single dose IV infusion of TY027 as compared to placebo up to Day 28
Proportion of COVID-19 patients tested negative for SARS-CoV-2 via reverse transcriptase-polymerase chain reaction (RT-PCR) | Up to Day 28
  Proportion of COVID-19 patients tested negative for SARS-CoV-2 via reverse transcriptase-polymerase chain reaction (RT-PCR) at Day 3, Day 5, Day 7, Day 14 and Day 28 after a single dose IV infusion of TY027 as compared to placebo
Proportion of COVID-19 patients with a minimum of 0.5 log time-weighted viral load reduction from saliva samples, via sub-genomic qRT-PCR | Day 7 post-dose or day of discharge, whichever is earlier
  Proportion of COVID-19 patients with a minimum of 0.5 log time-weighted viral load reduction from saliva samples, via sub-genomic qRT-PCR, at Day 7 post-dose or day of discharge, whichever is earlier, as compared to baseline between study groups

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Low, MBBS, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343